CLINICAL TRIAL: NCT06148246
Title: Family Fit: Promoting Family-Based Physical Activity and Weight Gain Prevention Through Mobile Technology
Brief Title: Family Fit Iterative App Development
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB202401844; R21HD100743 (NIH); IRB202102295 (Other: UF IRB)
Record Dates: First submitted 2023-11-17; First posted 2023-11-28 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Weight Gain Prevention; Physical Inactivity
Keywords: family-based; physical activity; exercise; mobile technology; wearables
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family Fit Condition (Intervention) (Experimental)
  Interventions: Behavioral: Family Fit Condition

INTERVENTIONS:
Behavioral: Family Fit Condition — Dyads in the Family Fit condition will use the Family Fit app and a Fitbit for 12 weeks, working to increase their moderate- to vigorous-intensity physical activity.

SUMMARY:
The overall aim of this study is to test the acceptability and usability of a mobile application (app) for family-based physical activity and weight gain prevention among parent/guardian and child (ages 9-12 years) dyads.

DETAILED DESCRIPTION:
This study includes a 12-week active intervention period. Interested participants will complete a study orientation webinar, then continue to a baseline visit and online questionnaires if interested. They will then complete 7-days of accelerometry monitoring to measure current physical activity levels. If eligible, they will attend a brief kick-off meeting to receive their Fitbits and study apps. The intervention period is 12 weeks, all remotely delivered. The intervention focuses on families working to increase their moderate- to-vigorous intensity physical activity. At 12 weeks, families will attend a brief in-person assessment visit and complete online questionnaires and 7 days of accelerometry, and complete a semi-structured interview via Zoom to discuss their experiences and provide feedback for future program modifications.

ELIGIBILITY:
Inclusion Criteria:

1. Parent (or legal guardian) must:

   * Be between 18-65 years old
   * Use a mobile Apple or Android device (e.g., smartphone, tablet)
   * Have a mobile data plan or reliable access to home Wi-Fi
   * Have an active Facebook account
2. Child must:

   * Be 9-12 years old
   * Live in the residence of parent (at least 50% of the time)
3. Child and parent must:

   * Be able to speak and read English.
   * Be insufficiently physically active (adult: <150 minutes/week moderate physical activity or <75 minutes/week vigorous physical activity, child: <6 days/week of 60 minutes moderate- to vigorous-intensity physical activity)
   * Be able to engage in physical activity.
   * Live within 75 miles of the UF campus

Exclusion Criteria:

1. Parent currently, or trying to become, pregnant.
2. Current participation in a structured physical activity or weight loss program (children playing sports will be permitted)
3. Currently enrolled in a research study focused on changing diet or physical activity.
4. Use of weight loss medications
5. Child current use of Fitbit (or similar physical activity device)
6. History of eating disorder
7. One parent and one child per family unit may enroll

Ages: 9 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-18 (Actual); Primary Completion 2025-07-06 (Actual); Study Completion 2025-07-16 (Actual)

PRIMARY OUTCOMES:
Recruitment | Baseline
  Number of dyads screened and enrolled; rate of recruitment
Use rates | 12 weeks
  Use rates of the Family Fit app summarized from back-end data from the app
Acceptability | 12 weeks
  Satisfaction, perceived appropriateness, intent to continue to use intervention materials, likelihood of recommending the program to a friend, open-ended questions: overall satisfaction with program and suggestions for improvement
Retention | 12 weeks
  Number of dyads per condition who complete follow-up assessments

SECONDARY OUTCOMES:
Sustainability | 12 weeks
  Use of Family Fit app, Fitbit app, and Fitbit devices from weeks 13-18
Usability | 12 weeks
  Scores from System Usability Scale
Contamination | 12 weeks
  Use of outside physical activity programs, devices, and apps during the study
Average minutes/day of moderate- to vigorous-intensity physical activity, accelerometry | Baseline, 12 weeks
  Actigraph accelerometers to be used; 7 days of wear time will be requested from participants at each time point
Average minutes/day of moderate- to vigorous-intensity physical activity, self-report | Baseline, 12 weeks
  Godin Leisure-Time Exercise Questionnaire
BMI (parents) | Baseline, 12 weeks
  Body weight (to the nearest 0.1 lbs), height (to the nearest 0.25 inch) with standard protocols; BMI calculated as kg/m^2
BMI percentile (child) | Baseline, 12 weeks
  Body weight (to the nearest 0.1 lbs), height (to the nearest 0.25 inch) with standard protocols; BMI percentile using standardized charts
Family cohesion | Baseline, 12 weeks
  Moos et al. family environment scale
Social support | Baseline, 12 weeks
  Kiernan et al. adaptation of social support scale
Family communication | Baseline, 12 weeks
  Measure from the National Longitudinal Study of Adolescent Health (Add Health)
Family engagement | Baseline, 12 weeks
  Measure from the National Longitudinal Study of Adolescent Health (Add Health)
Family closeness | Baseline, 12 weeks
  Measure from the National Longitudinal Study of Adolescent Health (Add Health)

CONTACTS AND LOCATIONS:
Overall Officials: Danielle E Jake-Schoffman, PhD, Principal Investigator — University of Florida
Locations (1):
- UF College of Health and Human Performance, Gainesville, Florida, United States

DOCUMENTS (1):
  • Informed Consent Form (2025-01-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT06148246/ICF_000.pdf